CLINICAL TRIAL: NCT01995994
Title: Continuous Glucose Monitoring System in Intensive Care Unit - Preliminary Study Evaluating Accuracy
Brief Title: Continuous Glucose Monitoring System in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Assistant Professor, Seoul National University Hospital
Other Study IDs: D-1203-106-404
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2013-11

CONDITIONS: Diabetic Blood Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RT-CGM

SUMMARY:
To assess the accuracy, safety, and influence of sampling site of Real-time continuous glucose monitoring system (Medtronic Guardian).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Staying in intensive care units longer than 72 hours

Exclusion Criteria:

* Skin disease
* DIC
* Immune suppressed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned to stay in intensive care units longer than 72 hours
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Difference between finger stick blood glucose and real-time continuous glucose monitoring | 72 hours

SECONDARY OUTCOMES:
Measurement error of real-time continuous glucose monitoring | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea